CLINICAL TRIAL: NCT05584644
Title: Treatment Patterns and Clinical Outcomes Among Indian Patients Receiving Palbociclib Combinations for HR+/HER2- Advanced/Metastatic Breast Cancer in Real World Settings
Brief Title: A Study to Describe the Breast Cancer Patient Population, Treatment, and Results in Indian Patients Receiving Combinations of the Medicines Called Palbociclib for Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481145
Record Dates: First submitted 2022-05-23; First posted 2022-10-18 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Breast Carcinoma; Breast Neoplasms; Breast Tumors; Cancer of Breast
Keywords: Hormone receptor positive / human epidermal growth factor 2 negative (HR+/HER2-); Advanced Breast Cancer; Metastatic Breast Cancer; Palbociclib; aromatase inhibitor; fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Palbociclib plus hormonal treatment - first line treatment: Patients who initiated Palbociclib + hormonal therapy in the first line treatment
  Interventions: Drug: Palbociclib plus hormonal treatment - first line treatment
- Palbociclib plus hormonal treatment - second line treatment: Patients who initiated palbociclib plus hormonal treatment in the second line treatment
  Interventions: Drug: Palbociclib plus hormonal treatment - second line treatment

INTERVENTIONS:
Drug: Palbociclib plus hormonal treatment - first line treatment — Palbociclib plus hormonal treatment
  Groups: Palbociclib plus hormonal treatment - first line treatment
Drug: Palbociclib plus hormonal treatment - second line treatment — Palbociclib plus hormonal treatment
  Groups: Palbociclib plus hormonal treatment - second line treatment

SUMMARY:
The purpose of this clinical study is to describe the patient population, breast cancer treatment, and breast cancer treatment results of adult female patients who have received palbociclib combination treatments for advanced or metastatic breast cancer in India.

There are two groups of patients this study will describe. The first group of patients will have received palbociclib in combination with aromatase inhibitor (as prescribed by the Physician) for the treatment of postmenopausal women with HR+/HER2- advanced breast cancer as initial endocrine-based therapy for their metastatic disease. The second group of patients will have received palbociclib for the treatment of hormone receptor HR+/HER2- advanced or metastatic breast cancer in combination with fulvestrant in women with disease progression following endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* HR+/HER2- breast cancer diagnosis with confirmed metastatic or advanced disease
* Received palbociclib with aromatase inhibitor (as prescribed by the Physician) as initial endocrine therapy in postmenopausal metastatic breast cancer (MBC) patients or with fulvestrant in patients who have progressed on prior endocrine therapy
* Patients on Leutinizing Hormone Releasing Hormone (LHRH) agonists for ovarian function suppression in pre- or perimenopausal stage only if prescribed palbociclib with fulvestrant
* No prior or current enrolment in an interventional clinical trial for advanced/metastatic breast cancer
* Minimum of 3 months of follow up data since palbociclib with fulvestrant initiation, or minimum of 6 months of follow up data since palbociclib with aromatase inhibitor initiation

Exclusion Criteria:

* Cancers other than breast cancer
* Male breast cancer
* Visceral crisis

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult menopausal women with confirmed metastatic or advanced breast cancer in India
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- India (6):
  - Hemato Oncology Clinic Ahmedabad Private Limited, Rajpath Club Lane ,Gujarat, India, Ahmedabad
  - Max Super Speciality Hospital, Patparganj, Delhi, India
  - HCG Cancer Centre, Ahmedabad, Gujarat, India
  - Indo-American Hospital, Nandi Nagar, Banjara Hills, Hyderabad, Telangana, India
  - Bhagwan Mahaveer Cancer Hospital and Research Centre, Bajājnagar, Jaipur, Rajasthan, India
  - Max Super Speciality Hospital, Saket Institutional Area,, Saket, NEW Delhi, India

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with hormone receptor positive (HR+) /human epidermal growth factor receptor 2 negative (HER2-) advanced/metastatic breast cancer (ABC/MBC), who received palbociclib combined with aromatase inhibitor in menopausal state as initial endocrine therapy in MBC or with fulvestrant after progression on prior endocrine therapy were observed.
Pre-assignment Details: This retrospective observational study used medical records of participants from 6 oncology hospitals within a period of Dec 2016 to May 2021 (approximately 4.5 years). Available data was evaluated in 9 months of this retrospective observational study.
Groups:
- Palbociclib: 1st Line Therapy: Participants who received palbociclib in combination with hormonal therapy as first line therapy under standard real world practice for HR+/HER2- MBC were included in this retrospective observational study. Available data were evaluated in 9 months of this study.
- Palbociclib: 2nd Line Therapy: Participants who received palbociclib in combination with hormonal therapy as second line therapy under standard real world practice for HR+/HER2- MBC were included in this retrospective observational study. Available data were evaluated in 9 months of this study.
Period: Overall Study
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Started | 105 | 45
Completed | 105 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy | Total
Number analyzed (Participants) | 105 | 45 | 150
Age, Customized [Count of Participants; unit: Participants]
  Less than or equal to (<=) 65 years | 66 | 32 | 98
  Greater than (>) 65 years | 39 | 13 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 45 | 150
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to the Starting Dose of Palbociclib
Description: Number of participants according to their starting dose (125 milligrams per day [mg/day], 100 mg/day) of palbociclib were reported in this outcome measure. For participants whose dose details were not available was reported under 'data not available'. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: From index date until end of follow-up (anytime from Dec 2016 to May 2021[approximately 4.5 years]); available data studied from 24-May-2021 to 22-Feb-2022 (approximately 9 months of this study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  125mg/day | 99 | 43
  100mg/day | 1 | 2
  Data not available | 5 | 0

2. Primary Outcome: Duration of Treatment
Description: Duration of treatment was reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: From index date to end of treatment, from Dec 2016 to May 2021 (approximately 4.5 years); available data studied from 24-May-2021 to 22-Feb-2022 (approximately 9 months of this study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Months | 15.08 [9.67 to 22.43] | 11.63 [6.37 to 19.60]

3. Primary Outcome: Number of Participants Who Had Any Palbociclib Dose Reduction
Description: Number of participants according to dose reductions during palbociclib treatment were reported in this outcome measure. Dose was reduced to 100mg and 75 mg. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Dose reduced to 100 mg | 13 | 1
  Dose reduced to 75 mg | 1 | 0

4. Primary Outcome: Number of Participants Who Had Any Interruption in Palbociclib Treatment
Description: Number of participants with any interruptions during palbociclib treatment were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants | 9 | 1

5. Primary Outcome: Number of Participants Who Had Any Delays in Palbociclib Treatment
Description: Number of participants who had any delay in palbociclib treatment were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants | 7 | 1

6. Primary Outcome: Number of Participants According to Reasons for Treatment Discontinuation
Description: Number of participants classified according to reasons for treatment discontinuations which included increased transaminases, cardiomyopathy was reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Increased transaminases | 1 | 0
  Cardiomyopathy | 1 | 0

7. Primary Outcome: Number of Participants According to Reasons for Change in Treatment
Description: Number of participants classified according to reasons for change in treatment were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 18 | 18
Participants
  Side effects/toxicity | 10 | 3
  Other reasons | 5 | 0
  Dose Reduced | 12 | 4
  Dose Resumed following interruption or cycle delay | 9 | 3
  Dose Interrupted (temporarily stopped during a dose cycle) | 9 | 1
  Cycle delay (the next cycle is pushed back) | 7 | 1
  Combination partner therapy continued | 17 | 3

8. Primary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from palbociclib combination treatment initiation until 1) clinician documented disease progression (PD) while on palbociclib, 2) death, 3) start of a new therapy line after final palbociclib dose, if the reason for discontinuation of palbociclib was disease progression, or 4) last available follow-up, whichever occurred first. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: From index date to death or disease progression start of new therapy or last available follow-up whichever occurred first,maximum up to approximately 4.5years;available data studied from 24-May-2021 to 22-Feb-2022 (approximately 9 months of this study)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 77 | 28
Months | 31.97 [22.43 to 47.50] | 22.33 [11.80 to 48.80]

9. Primary Outcome: Objective Response Rate (ORR)
Description: The objective response rate was defined as the percentage of participants with complete response (CR) and partial response (PR). As per RECIST version 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); PR = at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: From index date to CR/PR, from Dec 2016 to May 2021 (approximately 4.5 years); available data studied from 24-May-2021 to 22-Feb-2022 (approximately 9 months of this study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Percentage of participants | 63.81 | 77.78

10. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: From index date to death, from Dec 2016 to May 2021 (approximately 4.5 years); available data studied from 24-May-2021 to 22-Feb-2022 (approximately 9 months of this study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants | 8 | 3

11. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from index date to the date of death due to any cause. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: From index date to death due to any cause, (from Dec 2016 to May 2021 [approximately 4.5 years]); available data studied from 24-May-2021 to 22-Feb-2022 (approximately 9 months of this study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Months | NA [NA to NA] — Median and 95%CI could not be calculated as there were less number of participants with event. | NA [NA to NA] — Median and 95%CI could not be calculated as there were less number of participants with event.

12. Primary Outcome: Number of Participants According to Biomarker Status
Description: Number of participants classified according to the biomarker status were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants | NA — The data of eligible participants were not available on medical records. | NA — The data of eligible participants were not available on medical records.

13. Primary Outcome: Number of Participants With Family History of Breast Cancer
Description: Number of participants with family history of breast cancer were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants | 4 | 0

14. Primary Outcome: Duration From Breast Cancer Diagnosis to Palbociclib Treatment
Description: Duration from breast cancer diagnosis to palbociclib treatment was reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Months | 8.69 (26.12) | 45.50 (43.53)

15. Primary Outcome: Number of Participants According to Stages of Breast Cancer
Description: Number of participants classified according to stages (Stage I, II, IIIa, IV) of breast cancer were included in this outcome measure. Stage I indicated the cancer was small and had not spread anywhere else, Stage II indicated the cancer had grown, but had not spread, Stage IIIa indicated the cancer had grown larger and might have spread to the surrounding tissues and/or the lymph nodes. Stage IV indicated the cancer had spread from where it started to at least 1 other body organ, also known as secondary or metastatic cancer. For participants whose breast cancer stage were not available was reported under 'data not available'. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Stage I | 5 | 0
  Stage II | 5 | 12
  Stage IIIa | 1 | 1
  Stage IV | 70 | 31
  Data not available | 24 | 1

16. Primary Outcome: Number of Participants According to Node Status
Description: Number of participants classified according to node status were included in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Distal | 6 | 1
  Regional nodes | 5 | 5

17. Primary Outcome: Number of Participants According to Menopausal Status
Description: Number of participants classified according to menopausal status which included natural and induced were included in this outcome measure. For participants whose details were not available was reported under 'data not available'. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Induced | 16 | 16
  Natural | 88 | 29
  Data not available | 1 | 0

18. Primary Outcome: Number of Participants According to Performance Status Based on Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG PS was used to assess physical health of participants. ECOG PS grade:0= fully active, able to carry on all pre-disease performance without restriction,1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature 2= ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours, 3= capable of only limited self-care, 4= completely disabled, cannot carry on any selfcare totally confined to bed or chair confined to bed or chair more than 50% of waking hours and 5= dead. Participants whose ECOG scores were not available reported as 'data not available'. Only those categories with non-zero values were reported. Index date= 60 days after physician first prescribed palbociclib + hormonal following availability of specific indication in market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  1 | 65 | 33
  2 | 6 | 5
  3 | 0 | 1
  Data not available | 34 | 6

19. Primary Outcome: Number of Participants According to Metastatic Sites
Description: Number of participants classified according to metastatic sites were reported in this outcome measure. Metastatic sites included bone, lung, liver, lymph nodes, others. For participants whose details were not available was reported under 'data not available'. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market. Participant could have more than 1 location of metastases.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Bone | 62 | 28
  Lung | 28 | 16
  Liver | 14 | 7
  Lymph nodes | 16 | 6
  Others | 7 | 4
  Data not available | 12 | 3

20. Primary Outcome: Number of Participants According to de Novo and Recurrent Disease
Description: Participants classified according to status of disease as de novo versus and recurrent disease were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants | NA — The data of eligible participants were not available on medical records. | NA — The data of eligible participants were not available on medical records.

21. Primary Outcome: Number of Participants According to Therapies Received for Early Breast Cancer
Description: Participants classified according to therapies received for early breast cancer which included adjuvant chemotherapy, adjuvant endocrine therapy, neoadjuvant treatment, radiotherapy, surgery were reported in this outcome measure. For participants whose details were not available was reported under 'data not available'. Participant could have received more than 1 therapy. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Adjuvant chemotherapy | 4 | 8
  Adjuvant endocrine therapy | 14 | 5
  Neoadjuvant treatment | 6 | 11
  Radiotherapy | 20 | 26
  Surgery | 13 | 26
  Data not available | 69 | 9

22. Primary Outcome: Time Since End of Adjuvant Treatment
Description: Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Months | NA [NA to NA] — The data of eligible participants were not available on medical records. | NA [NA to NA] — The data of eligible participants were not available on medical records.

23. Primary Outcome: Number of Participants According to Supportive Therapies Received for Hormone Receptor Positive / Human Epidermal Growth Factor 2 Negative (HR+/HER2-) Diagnosis
Description: Participants were classified according to supportive therapies received for HR+/HER2- diagnosis and were reported in this outcome measure. Supportive therapies included nutritional treatment, bisphosphonates, anti-anxiety, anti-depressant, anti-emetics, non-steroidal anti-inflammatory drugs. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants
  Nutritional support | 37 | 7
  Bisphosphonates | 8 | 2
  Antibiotics | 5 | 1
  Anti-anxiety | 3 | 0
  Anti-depressants | 1 | 0
  Anti-emetics | 1 | 1
  Opioid extended release | 1 | 0
  Opioid immediate release | 1 | 0
  Non-steroidal anti-inflammatory drugs | 1 | 0
  Other supportive care | 36 | 3
  NA | 50 | 36

24. Primary Outcome: Duration of Supportive Treatments for ABC/MBC
Description: as for outcome 22
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Months | NA [NA to NA] — The data of eligible participants were not available on medical records. | NA [NA to NA] — The data of eligible participants were not available on medical records.

25. Primary Outcome: Number of Participants According to Reasons for Regimen Change
Description: Participants were classified according to reasons for regimen change and were reported in this outcome measure. Index date was defined as 60 days after the physician first prescribed palbociclib + hormonal therapy (letrozole, fulvestrant or anastrozole for first line and letrozole, fulvestrant or exemestane for second line therapy) following the availability of specific indication in the market.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
Number analyzed (Participants) | 105 | 45
Participants | NA — The data of eligible participants were not available on medical records. | NA — The data of eligible participants were not available on medical records.

ADVERSE EVENTS:
Time Frame: From index date until end of follow up (anytime from Dec 2016 to May 2021[approximately 4.5 years]); available data studied from 24-May-2021 to 22-Feb-2022 (approximately 9 months of this study)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Palbociclib: 1st Line Therapy | Palbociclib: 2nd Line Therapy
All-Cause Mortality (participants affected / at risk) | 8/105 | 3/45
Serious Adverse Events (participants affected / at risk) | 4/105 | 0/45
Other Adverse Events (participants affected / at risk) | 2/105 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib: 1st Line Therapy (N=105) | Palbociclib: 2nd Line Therapy (N=45)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Acute Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib: 1st Line Therapy (N=105) | Palbociclib: 2nd Line Therapy (N=45)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Increased Transaminases (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT05584644/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT05584644/SAP_001.pdf